CLINICAL TRIAL: NCT02567929
Title: Assessment of the Anesthetic Effect on the Activity of Immune Cell in Patient With Breast Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Konkuk University Medical Center (Other)
Responsible Party: Principal Investigator, Seong-Hyop Kim, Associate Professor, Konkuk University Medical Center
Allocation: Randomized | Model: Factorial | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: KUH1160086
Record Dates: First submitted 2015-09-02; First posted 2015-10-05 (Estimated); Last update posted 2018-04-02 (Actual); Status verified 2018-03

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Propofol; Sevoflurane

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- propofol group (Active Comparator): The patient who anesthetized by using propofol.
  Interventions: Drug: propofol group
- sevoflurane group (Active Comparator): The patient who anesthetized by using propofol
  Interventions: Drug: sevoflurane group

INTERVENTIONS:
Drug: propofol group — Patient will be anesthetized by using propofol infusion during operation.
  Other Names: propofol
  Arms: propofol group
Drug: sevoflurane group — Patient will be anesthetized by using sevoflurane inhalation during operation.
  Other Names: sevoflurane
  Arms: sevoflurane group

SUMMARY:
Anesthetics agents has variety inflammation during the cancer surgery. This perioperative inflammation can influence to cancer metastasis or recurrence.

The purpose of this study is to prove the variation of immune cell activity between preoperative and postoperative period.

DETAILED DESCRIPTION:
The patients were allocated randomly to receive propofol or sevoflurane. Also, a total of 18ml of blood sample was obtained for total 3 times in consecutive order.

1. immediate before anesthesia induction
2. postoperative 1 hours
3. postoperative 24 hours

Serum in blood will be obtained and activity of helper T cell, natural killer cell and level of serum cytokine will be evaluated by flow cytometry or enzyme-linked immunosorbent assay

ELIGIBILITY:
Inclusion Criteria:

* patient who was planned to undergo colon cancer surgery.

Exclusion Criteria:

* age < 20 years old
* history of hypersensitivity reaction in propofol or sevoflurane
* history of previous cancer
* patient with ongoing inflammation

Min Age: 20 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 218 (Actual)
Dates: Start 2016-03 (Actual); Primary Completion 2016-12 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
CD39 and CD73 on circulating regualtory T cells | preoperative time. postoperative 1 hours and 24 hours
  change of percentage of CD39 and CD73 (scores range from 0 to 100)

SECONDARY OUTCOMES:
Circulating natural killer cells | preoperative time. postoperative 1 hours and 24 hours
  change of percentage of circulating natural killer cell (scores range from 0 to 100)

OTHER OUTCOMES:
Circulating type 1 and type 17 helper T cells | preoperative time. postoperative 1 hours and 24 hours
  change of percentage of helper T cell (scores range from 0 to 100)

CONTACTS AND LOCATIONS:
Overall Officials: Seong-Hyop Kim, M.D,Ph.D, Principal Investigator — Konkuk University Medical Center
Locations (1):
- Konkuk University Medical Center, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No